CLINICAL TRIAL: NCT06759428
Title: Registry of Chronic Subdural Hematoma
Acronym: CSDH Registry
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, R. Dammers, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2021-0629
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Chronic Subdural Hematoma; Registry
Keywords: Chronic subdural hematoma; Traumatic Brain Injury; Registry; Treatment outcome; Burr hole drainage; modified Rankin Scale
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CSDH patients: All adult patients diagnosed with chronic subdural hematoma who provide informed consent to participate in the study will be included. Participants will receive standard care, with treatment determined by their treating physician based on clinical judgment. Treatment options may include burr hole drainage, craniotomy, embolization of the middle meningeal artery, pharmacological management, or a wait-and-scan approach. Follow-up will be conducted at 3 months via a telephone interview.

SUMMARY:
The goal of this observational study is to better understand how chronic subdural hematoma (CSDH) progresses and how patients are treated and cared for. The study focuses on three main questions:

1. What are the characteristics of patients with CSDH when they are diagnosed?
2. What treatments do patients with CSDH receive?
3. What are the outcomes for patients with CSDH, including their functional ability, cognitive health, and neurological status?

Participants will receive their usual standard treatment. As part of the study, they will complete a brief telephone interview three months after their treatment.

DETAILED DESCRIPTION:
Rationale:

Chronic subdural hematoma (CSDH) is a common condition encountered by neurologists and neurosurgeons. While guidelines for the management of CSDH have recently been developed, high-quality evidence to inform these recommendations, particularly level I evidence from randomized clinical trials (RCTs), is awaited. Significant variability in the management of CSDH persists at international, national, and inter-hospital levels. To further refine and implement evidence-based guidelines, a detailed understanding of current clinical practices and their associated outcomes is essential.

Objective:

To describe the baseline characteristics, treatment strategies, and outcomes of patients diagnosed with chronic subdural hematoma.

Study design:

A prospective, observational multicenter cohort study.

Study population:

All adult patients diagnosed with chronic subdural hematoma.

Main study parameters/endpoints:

The primary endpoint is functional outcome, measured by the modified Rankin Scale (mRS) at 3 months. Secondary endpoints, also assessed at 3 months, include recurrence, mortality, complications, hospital length of stay, Markwalder Grading Scale (MGS), modified National Institutes of Health Stroke Scale (mNIHSS), and Telephone Interview for Cognitive Status (TICS).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients will be treated in accordance with standard clinical practice. Study participation imposes minimal additional burden, consisting of a single telephone interview at three months, estimated to take approximately 10 minutes. The findings from this registry are expected to benefit future CSDH patients by informing evidence-based guidelines and improving care practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CSDH
* 18 years or older

Exclusion Criteria:

* Patients who do not consent to participate in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with CSDH will be recruited from participating centers.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score at 3 months following diagnosis | 3 months following diagnosis
  Functional outcome assessed using the modified Rankin Scale (mRS), a 6-point scale where 0 indicates no symptoms, higher scores reflect greater disability, and 6 represents death.

SECONDARY OUTCOMES:
Recurrence rate within 3 months following diagnosis | 3 months following diagnosis
  Recurrence of symptoms following initial, persistent improvement, confirmed by imaging as CSDH, and potentially requiring reoperation.
Mortality within 3 months following diagnosis | 3 months following diagnosis
  All-cause mortality.
Complications within 3 months following diagnosis | 3 months following diagnosis
  Complications after treatment of CSDH.
Duration of hospital stay | 3 months following diagnosis
  Total number of days admitted to the hospital for CSDH-related causes.
Markwalder Grading Scale (MGS) score at 3 months following diagnosis | 3 months following diagnosis
  Neurological outcome assessed using the Markwalder Grading Scale (MGS), a 4-point scale where 0 indicates no symptoms, higher scores reflect greater neurological disability, and 4 represents coma.
modified National Institutes of Health Stroke Scale (mNIHSS) score at 3 months following diagnosis | 3 months following diagnosis
  Neurological outcome assessed using the modified National Institutes of Health Stroke Scale (mNIHSS), a standardized tool ranging from 0 to 31, where 0 indicates no neurological deficits, and higher scores reflect increasing severity of stroke-related impairments.
Telephone Interview for Cognitive Status (TICS) score at 3 months following diagnosis | 3 months following diagnosis
  Cognitive status assessed using the Telephone Interview for Cognitive Status (TICS), a standardized tool ranging from 0 to 50, where higher scores indicate better cognitive functioning, and lower scores reflect greater cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Dammers, Principal Investigator — Erasmus Medical Center; Dagmar Verbaan, Principal Investigator — Amsterdam UMC
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
De-identified research data may be shared with third parties to enhance its scientific value. Requests for data must be submitted to the principal investigators, accompanied by a detailed description of the study's objectives and methods. Data will be available for sharing beginning in January 2028. Sharing will be permitted for scientific purposes, such as individual patient meta-analyses. Additionally, explicit consent will be required for sharing de-identified data outside the European Union.
Time Frame: Data will be available for sharing beginning in January 2028.
Access Criteria: Written proposals will be reviewed by the registry's principal investigators to evaluate their suitability for data use. Before any data is shared, a data-sharing agreement compliant with Dutch regulations will be established.

REFERENCES:
- See also: This link provides access to the official website of the study, offering a description of the project, including its objectives, methodology, and relevant details. — https://www.dshr.one/registry